CLINICAL TRIAL: NCT00703612
Title: Phase I/II Study of Intravenous Administration of Activated Autologous Adipose-Derived Stromal Vascular Fraction in Patients With Type 2 Diabetes
Brief Title: Safety and Efficacy of Autologous Adipose-Derived Stem Cell Transplantation in Type 2 Diabetics
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Adistem Ltd (Industry)
Responsible Party: Bill Paspaliaris / Director, Adistem Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adis-002
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2008-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Adipose-derived stem cells; Adipose stromal vascular fraction; Autologous; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): This is the only arm and that is the treatment group.
  Interventions: Procedure: Autologous Adipose-derived Stem cells

INTERVENTIONS:
Procedure: Autologous Adipose-derived Stem cells — Intravenous administration of autologous activated stromal vascular fraction derived from 100-120 ml lipoaspirate following mini-liposuction of abdominal adipose tissue.

SUMMARY:
The purpose of this study is to determine whether intravenous administration of autologous adipose-derived stem cells is of benefit in the management of types 2 diabetics.

DETAILED DESCRIPTION:
Diabetes Mellitus is of large epidemic proportions worldwide. It is proliferating at such a fast rate that new novel drugs and other therapeutic approaches are required. The purpose of this Phase 1/Phase 2 study is to determine whether the intavenous administration of activated adipose-derived stromal vascular fraction as a single procedure is safe to and can benefit the disease pathology of patients with Type 2 Diabetes Mellitus (insulin resistance). Patients will be observed over 12 months following the procedure, with a 2 week, 1 month and then tri monthly diagnostics and life style questionaires.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Type II diabetes for at least 2 years
* Type 2 diabetics on oral hypoglycemic agents and/or insulin
* Fasting blood sugar of >200mg% on at least two occasions
* Willing to keep a weekly diary and undergo observation for 12 months

Exclusion Criteria:

* Presence of of previous and/or acute diabetic complications such as myocardial infarction, CVA or nephropathy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Lowering of blood glucose be it fasting, random or post prandial | At 2, 4, 12, 24, 36, and 48 weeks

SECONDARY OUTCOMES:
Decrease in anti-hyperglycemic medication dosages. | At 2, 4, 12, 24, 36, and 48 weeks.
Improvement in the general well-being of patients. | At 2, 4, 12, 24, 36, and 48 weeks.
Lowering of glycosylated hemoglobin (HbA1C). | At 4, 12, 24, 36, and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emeritta A Barrenechea, MD, Principal Investigator — Veterens Memorial Medical Centre, Philippines; Florencio Q Lucero, MD, Principal Investigator — University of Philippines, College of Medicine.; Letitia Lucero-Palma, MD, Study Director — Far Eastern University-NRMF Hospital, Quezon City, Philippines; Bill Paspaliaris, PhD, Study Chair — Adistem Ltd
Locations (2):
- Philippines (2):
  - Beverly Hills Medical Group, Makati City, Manila
  - Veterens Memorial Medical Centre, Quezon City, Manila

REFERENCES:
- [Background] Gimble JM, Katz AJ, Bunnell BA. Adipose-derived stem cells for regenerative medicine. Circ Res. 2007 May 11;100(9):1249-60. doi: 10.1161/01.RES.0000265074.83288.09. PMID 17495232